CLINICAL TRIAL: NCT01970423
Title: Central Sleep Apnea and New-onset Cardiac Resynchronization in Patients With Conventional Pacemaker or ICD Therapy: a Multicenter, Randomized Clinical Trial
Brief Title: Sleep Apnea and CRT Upgrading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Wolfgang Dichtl, MD PhD, Priv.-Doz. DDr., Medical University Innsbruck
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UPGRADE
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Cardiomyopathy
Keywords: Patients with pacemaker or ICD therapy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRT (Other): After randomization and polysomnography the CRT will get activated. After 3-5 months cross over to conventional right ventricular stimulation.
  Interventions: Device: CRT
- Right Ventricular Stimulation (Other): After randomization and polysomnography the conventional right ventricular stimulation will get activated. After 3-5 months cross over to CRT activation.
  Interventions: Device: conventional right ventricular stimulation

INTERVENTIONS:
Device: CRT — The new device is the first CRT-P that relies on a physiological parameter, respiration, to allow the pacemaker to follow the patient's breath and help create an appropriate pacing rate.
  Other Names: INLIVEN / VISIONIST (Boston Scientific); INCEPTA / AUTOGEN (Boston Scientific)
  Arms: CRT
Device: conventional right ventricular stimulation
  Arms: Right Ventricular Stimulation

SUMMARY:
Cardiac resynchronization therapy may reduce central sleep apnea, but there is no prospective randomized study so far demonstrating such an effect in patients with conventional pacemaker undergoing upgrading to CRT because of heart failure.

DETAILED DESCRIPTION:
Within the last decade cardiac resynchronization therapy (CRT) has been proven to be an effective therapy to reduce morbidity and mortality in chronic heart failure patients with wide QRS complex, in particular complete left bundle branch block. New indications have recently been established, including patients with mild symptoms and patients in need of conventional pacing such as high-grade atrioventricular block.

More than half - up to 80% - of patients with heart failure suffer from concomitant sleep apnea (SA), which further worsens symptoms and prognosis. Cardiac resynchronization therapy may ameliorate sleep apnea, but only the central form of sleep apnea (CSA). However, only very small uncontrolled studies with mainly less than 20 patients have been reported so far concerning the interactions between CRT and sleep apnea, and no data are available in patients with conventional right ventricular pacing undergoing upgrading to CRT.

Therefore, we want to perform a study called UPGRADE which is characterized

* being the first randomized study comparing the effects of new-onset cardiac resynchronization therapy on moderate and severe central sleep apnea, defined by an AHI ≥ 15/h as assessed by polysomnography in patients with conventional right ventricular pacing which is known to decrease cardiac function, induce heart failure and atrial fibrillation
* using a new technology called AP Scan® which enables continuous and reliable monitoring of sleep-disordered breathing (SDB); this technology is further validated with polysomnography, the gold standard in the diagnosis and follow-up in patients with sleep apnea

Unfortunately, one third of patients still do not benefit from CRT (so-called non-responders). On the other hand, up to 20% of patients greatly benefit and completely recover in terms of normalization of left ventricular ejection fraction and/or functional capacity (so-called super-responders). Research is urgently needed to decrease the number of non-responders and increase the number of super-responders.

Patient selection is still based on QRS duration and its morphology. Echocardiography and other imaging techniques for mechanical dyssynchrony assessment have failed to be a useful predictor for adequate patient selection. Therefore, we further want to test whether CRT itself does not only improve concomitant sleep apnea, but also if preexisting sleep apnea predicts the response to CRT in patients with previously conventional right-ventricular pacing undergoing an upgrade to CRT by additional implantation of a left ventricular lead.

ELIGIBILITY:
Inclusion Criteria:

* left ventricular ejection fraction < 50%
* implanted conventional pacemaker or ICD with a right ventricular pacing rate > 40% or planned "ablate and pace" therapy
* age 40 - 85 years

Exclusion Criteria:

* NYAH IV
* liver cirrhosis
* renal insufficiency (GFR < 30ml/min/1,73m²)
* expectancy of life < 1 year
* premenopausal woman
* drug or substance abuse
* hyperthyreosis
* custodianship
* CM allergy
* any condition that may compromise the compliance of the patient, or would preclude the patient from successful completion of the study
* plaster allergy
* enrollment in another clinical trial

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Improvement of central sleep apnea | January 2014 - June 2021
  improvement of moderate / severe central sleep apnea (AHI ≥ 15/h) due to new onset CRT as compared to ongoing conventional right ventricular pacing
Validation of the AP scan by the gold standard polysomnography | January 2014 - June 2021

SECONDARY OUTCOMES:
CRT response | January 2014 - June 2021
  secondary endpoints = CRT response according to pre-existing sleep apnea (RDI 0-14/h versus ≥ 15/h)
  * improvement of left ventricular ejection fraction and reduction in left ventricular endsystolic volume as assessed by transthoracic echocardiography
  * decrease in NTproBNP / BNP plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Dichtl, MD, Principal Investigator — Medical University of Innsbruck
Locations (2):
- Austria (2):
  - Medical University Innsbruck, Department for Internal Medicine III, Innsbruck
  - Medical University Innsbruck, Internal Medicine III (Cardiology & Angiology), Innsbruck